CLINICAL TRIAL: NCT04850196
Title: Effects of Transcutaneous Electrical Acupoint Stimulation on the Postoperative Sleep Quality and Postoperative Cognition in Elderly Patients Undergoing Laparoscopic Abdominal Surgery
Brief Title: TEAS on Sleep Quality and POCD in Elderly Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, principal investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TEAS and POCD
Record Dates: First submitted 2021-03-27; First posted 2021-04-20 (Actual); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Transcutaneous Electrical Acupoint Stimulation; Postoperative Sleep Disturbances; Postoperative Cognitive Dysfunction; Elderly Patients
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TEAS group (Experimental): TEAS treatment was performed for 30 mins before anesthesia on bilateral side by an experienced acupuncturist at the Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints And TEAS treatment for 30 mins was also performed on bilateral side by an experienced acupuncturist at the Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints at the end of surgery as well as on the each night before sleeping after surgery until discharged from the hospital
  Interventions: Device: TEAS
- Control group (Sham Comparator): Patients in the Control group received electrical stimulation at a non-acupoint which was located 2 cm interior to the bilateral Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints similar to patients in group TEAS.
  Interventions: Other: control group

INTERVENTIONS:
Device: TEAS — TEAS treatment was performed for 30 mins before anesthesia on bilateral side by an experienced acupuncturist at the Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints . And TEAS treatment for 30 mins was also performed on bilateral side by an experienced acupuncturist at the Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints at the end of surgery as well as on the each night before sleeping after surgery until discharged from the hospital
  Arms: TEAS group
Other: control group — Patients in the Control group received electrical stimulation at a non-acupoint which was located 2 cm interior to the bilateral Neiguan (PC6), HT7 (Shenmen), ST36 (Zusanli) and LI4 (Hegu) acupoints similar to patients in group TEAS
  Arms: Control group

SUMMARY:
Elderly patients are often considered as a high-risk population for major abdominal surgery due to reduced functional reserve and increased comorbidities. Previous study reported that about 40 and 10% of elderly (60 yr and older) patients suffered from postoperative cognitive dysfunction (POCD) 7 days and 3 months, respectively, after noncardiac surgery. POCD is a central nervous system complication after anesthesia and an operation, whose risk factors include age, education level, the operation (time, type, and mode), anesthesia (methods, drugs, and time) and postoperative analgesia. In the study of Su X et al, elderly patients are also more prone to develop postoperative sleep disturbances after surgery with prolonged sleep latencies, fragmented sleep, decreased sleep efficiency and abnormally sleep stages. Increasing evidence showed that sleep and circadian rhythm disturbances after surgery could promote β-amyloid peptide (Aβ) accumulation by simultaneously upregulating Aβ synthesis and interfering with Aβ clearance. This insoluble Aβ aggregates to form brain extracellular senile plaques, which are one of the neuropathological hallmarks of numerous postoperative cognitive disorders such as Alzheimer's disease(AD), and can be measured by amyloid positron emission tomography (PET) imaging through injecting 18F-florbetapir, a novel imaging agent that binds with high affinity (Kd 3.1 nM+0.7) to β-amyloid peptide fibrils in brain amyloid plaques, to the patients.Transcutaneous electrical acupoint stimulation (TEAS) is a new acupuncture therapy developed by combining transcutaneous electrical nerve stimulation (TENS) in European and American countries and traditional Chinese acupuncture. TEAS treat disease through inputting a pulse current of different frequencies, intensities, and waveforms via electrode paste adhering to the skin. Previous studies proved that TEAS has been successfully applied in many different procedures through stimulating different acupoints such as reducing postoperative pain, postoperative nausea and vomiting (PONV), and improving postoperative sleep quality. However, whether TEAS could affect Aβ deposition by improving postoperative sleep quality and thus affect the development of long-term cognitive impairment is still unclear. The aim of our study is to conduct the TEAS intervention to elderly patients who received laparoscopic abdominal surgery, and then to examine its effect on postoperative sleep quality, postoperative cognition and complications. In this study, we utilized 18F-florbetapir imaging to assess the relationships between postoperative sleep disturbances and POCD and brain Aβ burden through measuring by PET imaging.

ELIGIBILITY:
Inclusion Criteria:

* patient's age was 65 yr or older
* patient was scheduled to undergo elective major laparoscopic abdominal surgery (e.g., gastrointestinal and gynecologic surgery).
* the surgery was expected to last 2h or longer.

Exclusion Criteria:

* severe diseases in cardiovascular, respiratory, liver, kidney, or central nervous systems and having a life span of less than 3 months;
* a mini-mental status examination score (MMSE) of less than 23;
* a history of dementia or psychiatric illness;
* current use of sedatives, antidepressants or corticosteroids;
* alcoholism and drug dependence;
* difficulty with follow-up or poor compliance;
* patients with preoperative sleep disturbances;
* patients with sleep apnea or moderate and severe obstructive sleep apnea-hypopnea syndrome (OSAHS);
* patients with severe visual or hearing impairment or who were unable to communicate.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-04-10 (Estimated)

PRIMARY OUTCOMES:
Sleep Quality Assessment | on the first night before surgery (Preop 1)
  use the Athens Insomnia Scale (AIS): the total AIS scores range from 0 to 24 points with ≤ 4 indicating no combined with insomnia at night; 4-6 indicating suspicious insomnia at night; ≥ 6 points indicating a diagnosis of insomnia at night
Sleep Quality Assessment | the third night after surgery (POD 3).
  use the Athens Insomnia Scale (AIS): the total AIS scores range from 0 to 24 points with ≤ 4 indicating no combined with insomnia at night; 4-6 indicating suspicious insomnia at night; ≥ 6 points indicating a diagnosis of insomnia at night
Sleep Quality Assessment | the first week after surgery (POD 1W).
  use the Athens Insomnia Scale (AIS): the total AIS scores range from 0 to 24 points with ≤ 4 indicating no combined with insomnia at night; 4-6 indicating suspicious insomnia at night; ≥ 6 points indicating a diagnosis of insomnia at night
Sleep Quality Assessment | the sixth months after surgery (POD 6M).
  use the Athens Insomnia Scale (AIS): the total AIS scores range from 0 to 24 points with ≤ 4 indicating no combined with insomnia at night; 4-6 indicating suspicious insomnia at night; ≥ 6 points indicating a diagnosis of insomnia at night
Cognitive Assessment | on the first night before surgery (Preop 1)
  MMSE is a 30-point questionnaire that is widely used to evaluate the severity of cognitive impairment in individuals with cognitive disorders. Score cutoffs for the MMSE are as follows: greater than or equal to 24 for normal cognition, between 19 and 23 for MCI, between 10 and 18 for moderate cognitive impairment, and less than or equal to 9 for severe cognitive impairment.
Cognitive Assessment | the third night after surgery (POD 3).
  MMSE is a 30-point questionnaire that is widely used to evaluate the severity of cognitive impairment in individuals with cognitive disorders. Score cutoffs for the MMSE are as follows: greater than or equal to 24 for normal cognition, between 19 and 23 for MCI, between 10 and 18 for moderate cognitive impairment, and less than or equal to 9 for severe cognitive impairment.
Cognitive Assessment | the first week after surgery ( POD 1W)
  MMSE is a 30-point questionnaire that is widely used to evaluate the severity of cognitive impairment in individuals with cognitive disorders. Score cutoffs for the MMSE are as follows: greater than or equal to 24 for normal cognition, between 19 and 23 for MCI, between 10 and 18 for moderate cognitive impairment, and less than or equal to 9 for severe cognitive impairment.
Cognitive Assessment | the sixth month after surgery (POD 6M).
  MMSE is a 30-point questionnaire that is widely used to evaluate the severity of cognitive impairment in individuals with cognitive disorders. Score cutoffs for the MMSE are as follows: greater than or equal to 24 for normal cognition, between 19 and 23 for MCI, between 10 and 18 for moderate cognitive impairment, and less than or equal to 9 for severe cognitive impairment.
Aβburden PET imaging | Aβ PET imaging was performed on the first week after surgery ( POD 1W)
  participants were injected intravenously with fluorine 18-labeled florbetaben tracer (Neuraceq; Piramel Imaging), and imaging was performed approximately 60 minutes later as per a standard protocol using PET-computed tomography.
Aβburden PET imaging | Aβ PET imaging was performed on the sixth month after surgery (POD 6M).
  participants were injected intravenously with fluorine 18-labeled florbetaben tracer (Neuraceq; Piramel Imaging), and imaging was performed approximately 60 minutes later as per a standard protocol using PET-computed tomography.

SECONDARY OUTCOMES:
Postoperative pain assessment | 24 hours after surgery
  pain scores were assessed on the visual analogue scale (VAS), where 0 indicates painlessness, and 10 indicates severe pain. The VAS score was measured at 2, 4, 6, and 24 hours postoperatively.
Postoperative adverse effects assessment | 24 hours after surgery
  adverse effects during 24 hours after surgery such as respiratory depression, bradycardia, nausea and vomiting, and dizzy were recorded and treated accordingly.

IPD SHARING:
Plan to Share IPD: No